CLINICAL TRIAL: NCT07353749
Title: Efficacy and Safety of Methylprednisolone in Preventing Adverse Cerebrovascular Events After Flow-Diverter Stent Implantation in Patients With Unruptured Intracranial Aneurysms: A Multicenter, Prospective, Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: Efficacy and Safety of Methylprednisolone After Flow-Diverter Stent Implantation in Unruptured Intracranial Aneurysms
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Duan Chuanzhi (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); Guangdong Provincial People's Hospital (Other); Beijing Tiantan Hospital (Other); First Affiliated Hospital of Chongqing Medical University (Other); The Affiliated Hospital Of Southwest Medical University (Other); Guangdong 999 Brain Hospital (Other); Eighth Affiliated Hospital, Sun Yat-sen University (Other); ZhuHai Hospital (Other); First Affiliated Hospital of Harbin Medical University (Other); Henan Provincial People's Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Second Affiliated Hospital of Nanchang University (Other); West China Hospital (Other); Shengjing Hospital (Other); Tongji Hospital (Other); Zunyi Medical College (Other); Qilu Hospital of Shandong University (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); The Third Affiliated Hospital of Southern Medical University (Other Government); Dongguan People's Hospital (Other Government); Shantou Central Hospital (Other); the Affiliated hospital of Guilin medical university, China (Unknown); Huizhou Third People's Hospital, Guangzhou Medical University (Other); Guangdong Provincial Hospital of Integrated Traditional Chinese and Western Medicine (Unknown); Qingyuan People's Hospital (Other); Guigang People's Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); First Affiliated Hospital of Jinan University (Other); Shenzhen People's Hospital (Other); Meizhou People's Hospital (Other); First People's Hospital of Foshan (Other)
Responsible Party: Sponsor-Investigator, Duan Chuanzhi, Professor, Zhujiang Hospital
Organization: Zhujiang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LC2025D035
Record Dates: First submitted 2026-01-06; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Unruptured Intracranial Aneurysms; Cerebrovascular Event; Hemorrhagic Stroke; Methylprednisolone; Flow Diverter
Keywords: Flow-diverter devices; Intracranial aneurysm; Methylprednisolone; Cerebrovascular Event
MeSH Terms: conditions — Hemorrhagic Stroke; Intracranial Aneurysm | interventions — Methylprednisolone

STUDY DESIGN:
Intervention Model Description: The subject numbers and corresponding medication numbers are permanently identified and unique for each successfully randomized patient. If any patients who have been successfully randomized do not receive the trial medication or cannot be reassigned to others, their medication and medication numbers will be invalidated by the medication administrator. To ensure blinding during the trial execution, unblinded personnel responsible for administering and configuring the trial drug must sign a confidentiality agreement. Investigators, other blinded investigators, subjects, and sponsors will not have access to any information regarding group assignment or related documents pertaining to the trial drug.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The subject numbers and corresponding medication numbers are permanently identified and unique for each successfully randomized patient. If any patients who have been successfully randomized do not receive the trial medication or cannot be reassigned to others, their medication and medication numbers will be invalidated by the medication administrator. To ensure blinding during the trial execution, unblinded personnel responsible for administering and configuring the trial drug must sign a confidentiality agreement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methylprednisolone Group (Experimental): Participants in this group will receive the investigational drug Methylprednisolone (injectable formulation) in addition to the standard therapy for flow-diverting device implantation. The specific administration regimen is as follows: Starting preoperatively on the day of surgery (Day 1), Methylprednisolone will be administered intravenously (IV drip at 40-60 drops per minute) once daily (qd) for 3 consecutive days. The dose is 2 mg per kilogram of body weight (with a maximum single daily dose not exceeding 160 mg), dissolved in normal saline.
  Interventions: Drug: Methylprednisolone (Injectable Form)
- Placebo Control Group (Placebo Comparator): Participants in this group will receive a placebo that is identical in appearance, volume, and mode of administration to the investigational drug, in addition to the identical standard therapy. Its administration regimen-including the start time, drip rate, duration, and treatment course-is fully matched to that of the Experimental Group to rigorously maintain the double.
  Interventions: Drug: Placebo Injection

INTERVENTIONS:
Drug: Methylprednisolone (Injectable Form) — This clinical study involves a perioperative pharmacological intervention using Methylprednisolone (Methylprednisolone Sodium Succinate for injection).
  The intervention is characterized by a weight-based, short-course intravenous regimen initiated preoperatively. The specific and distinguishing protocol is as follows:
  Drug & Form: Methylprednisolone Sodium Succinate, injectable formulation.
  Route & Method: Intravenous infusion, dissolved in normal saline, administered at a rate of 40-60 drops per minute.
  Dosing: 2 mg per kilogram of body weight per dose, with a maximum single dose not exceeding 160 mg.
  Timing & Duration: The regimen begins preoperatively on the day of surgery (Day 1). It is administered once daily (qd) for a total of 3 consecutive days.
  This protocol defines a distinct perioperative corticosteroid strategy aimed at modulating the inflammatory response associated with flow-diverting device implantation. It is an add-on therapy to the standard surgical and antiplat
  Arms: Methylprednisolone Group
Drug: Placebo Injection — The placebo intervention is characterized by a volume-matched, short-course intravenous regimen designed to be indistinguishable from the active drug in all aspects of administration except for the active pharmaceutical ingredient. The specific and distinguishing protocol is as follows:
  Drug & Form: Matched Placebo (0.9% Sodium Chloride Injection), provided in an identical injectable formulation.
  Route & Method: Intravenous infusion, administered at an identical rate of 40-60 drops per minute.
  Dosing: The infusion contains no active drug. The volume of each infusion is matched to the volume of the Methylprednisolone solution prepared for a participant of equivalent weight in the experimental group.
  Timing & Duration: The regimen begins preoperatively on the day of surgery (Day 1). It is administered once daily (qd) for a total of 3 consecutive days, precisely mirroring the active treatment schedule.
  Arms: Placebo Control Group

SUMMARY:
Study Title: Testing Methylprednisolone to Prevent Strokes After a Stent Procedure for Brain Aneurysms

What is the purpose of this study? This study aims to find out if a short course of a steroid medicine called methylprednisolone can help prevent strokes and other brain-related complications in patients who have a "flow diverter" stent placed to treat an unruptured brain aneurysm. The main goal is to see if this treatment reduces the combined number of new strokes (both clot-related and bleeding-related) or brain injury-related deaths within the first 30 days after the procedure.

Who can participate? Adults aged 18 or older with an unruptured brain aneurysm (size 3-25mm) who are scheduled to receive a flow-diverting stent and can provide informed consent may be eligible. Key reasons someone might not be able to join include: having multiple aneurysms needing quick treatment, being pregnant or breastfeeding, having a history of recent stroke, having active infections or stomach ulcers, having severe kidney disease, having very high/uncontrolled blood pressure or blood sugar, or already being on long-term steroid therapy.

What will happen in the study?

This is a multicenter, randomized, double-blind study. This means:

Participants will be randomly assigned (like flipping a coin) to one of two groups.

One group will receive methylprednisolone. The other group will receive a placebo (an inactive substance that looks identical).

Neither the participants nor their doctors will know which treatment is being given.

All participants will receive the standard care for the stent procedure and aftercare.

How long will the study last? The treatment period is short (around the time of the procedure). Participants will be closely monitored in the hospital and will have a follow-up visit around 30 days after the procedure to check their health status.

What will be measured? The researchers will mainly track whether participants have any stroke or brain injury-related death in the first 30 days. They will also check for other complications like bleeding, infections, and changes in daily function and quality of life. Safety will be monitored throughout.

How many people will take part? The study plans to enroll approximately 864 participants across multiple hospitals.

Study Dates:

The study is expected to start enrolling patients in January 2026 and finish in August 2027.

Who is organizing the study? This study is sponsored and led by Zhujiang Hospital, Southern Medical University.

DETAILED DESCRIPTION:
Title: A Study on the Efficacy and Safety of Methylprednisolone in Preventing Cerebrovascular Adverse Events after Flow-Diverting Device Implantation in Patients with Unruptured Intracranial Aneurysms-A Multicenter, Randomized, Double-Blind, Placebo-Controlled Clinical Trial

Sponsor: Zhujiang Hospital, Southern Medical University Leading Institution: Zhujiang Hospital, Southern Medical University

Research Objectives:

Primary Objective: To evaluate the efficacy of methylprednisolone treatment on the composite outcome of any new cerebrovascular adverse event and neurologic death within 30 days after flow-diverting device implantation in patients with unruptured intracranial aneurysms (IAs).

Secondary Objectives:

1. Incidence of any cerebrovascular adverse event (ischemic or hemorrhagic brain events) within 72 hours, 5 days, and 30 days post-operation.
2. Incidence of any ischemic brain event (ischemic stroke, in-stent thrombosis, urgent revascularization) within 72 hours, 5 days, and 30 days post-operation.
3. Incidence of any hemorrhagic brain event (intraparenchymal hemorrhage, subarachnoid hemorrhage, or subdural hematoma) within 72 hours, 5 days, and 30 days post-operation.
4. All-cause mortality within 30 days post-operation.
5. Proportion of patients with a modified Rankin Scale (mRS) score of 0-2 at 30 days post-operation.
6. Proportion of patients with an mRS score of 3-5 at 30 days post-operation.
7. Incidence of transient ischemic attack (TIA) within 72 hours post-operation.
8. EQ-5D score at 30 days post-operation.
9. Safety endpoint: Incidence of no new moderate or severe adverse events within 72 hours, 5 days, and 30 days post-operation.
10. Secondary safety endpoints:

    * Incidence of any intracranial hemorrhage within 72 hours post-medication.
    * Incidence of systemic bleeding complications (including gastrointestinal bleeding, systemic subcutaneous hemorrhage).
    * Incidence of non-hemorrhagic serious adverse events.
    * Incidence of gastrointestinal bleeding within 7 days post-operation.
    * Incidence of pulmonary infection during hospitalization.

Research Hypothesis: Methylprednisolone treatment can effectively reduce the incidence of cerebrovascular adverse events and neurologic death within 30 days after flow-diverting device implantation in patients with unruptured intracranial aneurysms.

Study Design: Multicenter, randomized, double-blind, placebo-controlled, parallel-group clinical trial.

Sample Size: The study is designed as randomized, double-blind, parallel, placebo-controlled. The primary outcome is the composite cerebrovascular event within 30 days post-implantation, defined as any new target vessel-related event: (1) ischemic stroke, (2) hemorrhagic stroke, (3) neurologic death.

Based on prior observational studies, the estimated primary outcome rate is 4.7% in the methylprednisolone group and 12.4% in the control group. With a two-sided significance level α=0.05 and power 1-β=0.80, the calculated sample size is approximately 203 per group. Accounting for a 5% dropout rate, 214 participants per group (428 total) are needed.

Adopting a more conservative estimate (methylprednisolone group: 6.0%, placebo group: 11.5%), the calculated sample size is approximately 410 per group. With a 5% dropout rate, 432 participants per group (864 total) are needed.

Study Population:

Diagnostic Criteria: Patients with unruptured intracranial aneurysms confirmed by CTA, MRA, or DSA.

Inclusion Criteria:

1. Age ≥ 18 years.
2. IA diagnosed by CTA, MRA, or DSA.
3. IA size between 3-25 mm.
4. Patient and/or legal representative understands the study purpose, volunteers to participate, and provides written informed consent.
5. Patients scheduled for flow-diverting device treatment.
6. Willing to undergo follow-up evaluations as per the study protocol.

Exclusion Criteria:

1. Patients with two or more multiple aneurysms requiring treatment within one month.
2. Women who are planning pregnancy, pregnant, or breastfeeding.
3. Pre-morbid mRS score ≥ 2.
4. Patients with systemic infectious diseases (latent/active), ulcerative colitis, diverticulitis, liver cirrhosis, myasthenia gravis, ocular herpes simplex; contraindications to corticosteroids such as active peptic ulcer, severe fungal infection.
5. Ruptured, recurrent, infectious, or dissecting aneurysms; patients with arteriovenous malformation, dural arteriovenous fistula, spinal dural arteriovenous fistula, moyamoya disease, etc.
6. Symptomatic cerebral vascular stenosis ≥ 70%.
7. History of stroke (intracerebral hemorrhage, cerebral infarction) within the past 30 days.
8. Planned for other surgical/interventional procedures within 30 days.
9. Severe comorbidities unsuitable for anesthesia or surgery (e.g., major cardiac, pulmonary, hepatic, splenic, renal diseases, atrial fibrillation, brain tumor, severe active infection, DIC, severe psychiatric history).
10. Inability to receive antiplatelet or anticoagulant therapy.
11. Allergy to methylprednisolone sodium succinate.
12. Long-term preoperative hormone therapy (≥1 week) for other conditions.
13. Concomitant use of hepatic enzyme-inducing drugs (e.g., barbiturates, rifampin, carbamazepine, phenytoin) or inhibitors (e.g., erythromycin, ketoconazole).
14. Chronic hemodialysis or severe renal insufficiency (GFR <30 ml/min or creatinine >220 μmol/L).
15. Uncontrolled hypertension (SBP >180 mmHg or DBP >110 mmHg despite medication).
16. Blood glucose <2.8 mmol/L or >22.2 mmol/L.
17. Vaccination within the past month or planned vaccination.
18. Unwilling or unable to comply with follow-up requirements.
19. Life expectancy <6 months due to any end-stage disease.
20. Participation in another clinical trial.

Main Interventions:

Experimental Group: Methylprednisolone treatment.

Control Group: Placebo treatment.

Follow-up: Within 24 hours post-surgery, within 72 hours post-surgery, at postoperative day 5/early discharge, and at 30±7 days.

Evaluation Indicators:

Primary Outcome: Incidence of the composite outcome of any new cerebrovascular adverse event and neurologic death within 30 days post-implantation.

Secondary Outcomes: Incidence rates as specified in objectives (2) through (17) above at the defined time points.

Statistical Methods:

For the primary outcome, a Log-binomial regression model will be the primary method to calculate the Risk Ratio (RR) and 95% CI. A multivariate model adjusting for baseline variables (gender, age, aneurysm location, blood pressure grade) will be used. If convergence fails, robust Poisson regression or logistic regression will be employed as alternatives. A two-sided p-value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* （1）Aged ≥ 18 years; （2）Diagnosed with intracranial aneurysm (IA) via CTA, MRA, or DSA;

  （3）IA size ranging from 3 to 25 mm;

  （4）The patient and/or their authorized representative can understand the study purpose, voluntarily participate, and sign the informed consent form;

  （5）Patients scheduled to receive flow diverter treatment;

  （6）Patients willing to complete follow-up evaluations in accordance with the clinical study protocol.

Exclusion Criteria:

* （1）Patients with two or more multiple aneurysms who require secondary treatment within one month; （2）Female patients who are planning to become pregnant, are pregnant, or are breastfeeding;

  （3）Pre-onset modified Rankin Scale (mRS) score ≥ 2;

  （4）Patients complicated with systemic infectious diseases (latent or active stage), ulcerative colitis, diverticulitis, liver cirrhosis, myasthenia gravis, or ocular herpes simplex; patients with contraindications to glucocorticoids, such as active peptic ulcer and severe fungal infection;

  （5）Ruptured aneurysms, recurrent aneurysms, infectious aneurysms, dissecting aneurysms; complicated with arteriovenous malformation, dural arteriovenous fistula, spinal dural arteriovenous fistula, moyamoya disease, etc.;

  （6）Patients with symptomatic cerebrovascular stenosis ≥ 70%;

  （7）Patients who have had a stroke (cerebral hemorrhage, cerebral infarction) within the past 30 days;

  （8）Patients scheduled to undergo other surgical/interventional procedures within 30 days;

  （9）Patients with severe comorbidities unsuitable for anesthesia or surgical treatment, such as major diseases of the heart, lungs, liver, spleen, and kidneys, atrial fibrillation, brain tumors, severe active infections, disseminated intravascular coagulation, and severe psychiatric history;

  （10）Patients who cannot receive antiplatelet aggregation or anticoagulant therapy;

  （11）Hypersensitivity to methylprednisolone sodium succinate;

  （12）Patients receiving long-term hormone therapy (≥ 1 week) due to other comorbidities before surgery;

  （13）Patients taking hepatic enzyme-inducing drugs, such as barbiturates, rifampicin, rifabutin, carbamazepine, phenytoin, primidone, and aminoglutethimide; or patients taking hepatic enzyme-inhibiting drugs, such as erythromycin and ketoconazole;

  （14）Patients undergoing chronic hemodialysis or with severe renal insufficiency (glomerular filtration rate < 30 ml/min or serum creatinine > 220 μmol/L (2.5 mg/dl));

  （15）Systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg that is uncontrollable with oral antihypertensive drugs;

  （16）Blood glucose < 2.8 mmol/L or > 22.2 mmol/L;

  （17）Patients who have received a vaccine injection within the past month or have a plan for vaccination;

  （18）Patients who cannot understand or are unwilling to complete follow-up evaluations in accordance with the clinical study protocol;

  （19）Patients with advanced diseases with an expected life expectancy of < 6 months;

  （20）Patients currently participating in other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 864 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of the Composite Outcome of Any New Cerebrovascular Adverse Event and Neurologic Death within 30 Days | From the implantation procedure (Day 1) up to 30 days post-procedure (assessed at visits V2 to V5).
  This primary efficacy endpoint measures the proportion of participants experiencing at least one of the following within 30 days post-implantation: a new ischemic event (ischemic stroke, stent thrombosis, or urgent revascularization), a new hemorrhagic event (any intracranial hemorrhage classified by the Heidelberg Bleeding Classification), or neurologic death. The outcome is calculated as the number of participants meeting this composite definition divided by the total participants in the group, multiplied by 100%.

SECONDARY OUTCOMES:
Incidence of Any Cerebrovascular Adverse Event | Within 72 hours (V2), at Postoperative Day 5 or early discharge (V3/V4), and within 30 days (V5).
  The proportion of participants with any new cerebrovascular adverse event (ischemic or hemorrhagic, as per primary outcome definitions) assessed at specific postoperative intervals.
Incidence of Any Ischemic Brain Event | Within 72 hours (V2), at Postoperative Day 5 or early discharge (V3/V4), and within 30 days (V5).
  The proportion of participants experiencing an ischemic brain event, including ischemic stroke, TIA, stent thrombosis, urgent revascularization, or cerebrovascular death.
Incidence of Any Hemorrhagic Brain Event | Within 72 hours (V2), at Postoperative Day 5 or early discharge (V3/V4), and within 30 days (V5).
  The proportion of participants experiencing a hemorrhagic brain event, defined as intraparenchymal hemorrhage, subarachnoid hemorrhage, or subdural hematoma.
Functional Outcome - mRS Score Distribution | At 30 days post-procedure (V5).
  The proportion of participants classified with favorable (mRS score 0-2) and unfavorable (mRS score 3-5) functional outcomes based on the modified Rankin Scale at 30 days.
Incidence of Transient Ischemic Attack (TIA) within 72 hours | Within 72 hours post-procedure (V2).
  The proportion of participants experiencing a TIA, characterized by transient neurological deficits without acute infarction on imaging.
Health-Related Quality of Life (EQ-5D) | At 30 days post-procedure (V5).
  The score derived from the EQ-5D descriptive system and Visual Analogue Scale (VAS), providing a utility index and a self-rated health assessment.
Safety Endpoint - Freedom from New Moderate/Severe Adverse Events | Within 72 hours (V2), at Postoperative Day 5 (V3), and within 30 days (V5).
  The proportion of participants who do not experience any new moderate or severe adverse event, including specific events like severe infections, new-onset diabetes, significant bleeding, fractures, or cardiovascular events.
Other Safety Endpoints | Various time frames as specified per endpoint, spanning from medication administration through the 30-day postoperative period and hospitalization.
  A series of safety measures assessing specific complications: intracranial hemorrhage within 72h post-medication; systemic bleeding complications; non-hemorrhagic serious adverse events; gastrointestinal bleeding within 7 days; and pulmonary infection during hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Chuanzhi Duan, Study Director — Southern Medical University, China
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided